CLINICAL TRIAL: NCT02358265
Title: A Multi-center, Randomized, Double Blind, Dose Escalating Phase III Study on the Efficacy, Safety and Long Term Outcome of Continuous vs. on Demand Treatment of Chronic Spontaneous Urticaria With Rupatadine.
Brief Title: Chronic Urticaria - Long Term Assessment of Effects of Rupatadine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, K. Weller, MD; PD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-LATER
Record Dates: First submitted 2014-12-18; First posted 2015-02-06 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — rupatadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mg Rupatadine on demand (Active Comparator): Rupatadine 10 mg, on demand
  Interventions: Drug: 10 mg Rupatadine on demand
- 10 mg Rupatadin (Active Comparator): Rupatadine 10 mg, continuously
  Interventions: Drug: 10 mg Rupatadine
- 20 mg Rupatadine (Active Comparator): Rupatadine 20 mg, continuously
  Interventions: Drug: 20 mg Rupatadine
- 10 mg rupatadine on demand (sham upd.) (Active Comparator): Rupatadine 10 mg, on demand (sham updosing to 20 mg)
  Interventions: Drug: 10 mg Rupatadine on demand (sham updosing to 20 mg)

INTERVENTIONS:
Drug: 10 mg Rupatadine on demand — Group A1 (dose administered: 10 mg rupatadine on demand): one tablet of placebo once daily- one on-demand tablet of rupatadine 10 mg intake only if needed.
  Arms: 10 mg Rupatadine on demand
Drug: 10 mg Rupatadine — Group B1 (dose administered: 10 mg rupatadine continuously): one tablet of rupatadine 10 mg once daily, one on-demand tablet of placebo, intake only if needed.
  Arms: 10 mg Rupatadin
Drug: 20 mg Rupatadine — Group B2 (dose administered: 10 mg rupatadine continuously): two tablets of rupatadine 10 mg daily- one on-demand tablet of placebo , intake only if needed.
  Arms: 20 mg Rupatadine
Drug: 10 mg Rupatadine on demand (sham updosing to 20 mg) — Group A2 (dose administered: 10 mg rupatadine on demand): two tablets of placebo daily- one on-demand tablet of rupatadine 10 mg ,intake only if needed.
  Arms: 10 mg rupatadine on demand (sham upd.)

SUMMARY:
To compare CSU disease activity at the end of the follow up phase between patients that had been treated daily continuously vs. on-demand in the treatment phase

DETAILED DESCRIPTION:
The treatment of CSU with nsAHs is currently the most common and only licensed therapeutic option to reduce the patients' wheal and flare type skin reactions and pruritus. CSU is a highly fluctuating disease and the severity of symptoms can change markedly from day to day. This is one of the reasons why, in routine daily practice, many patients tend to perform an on demand rather than a continuous, daily, preventive treatment of their symptoms with nsAHs. While in the field of allergic rhinitis several studies point towards a better efficacy of nsAHs if continuously given (6-8), the only study in CSU comparing both treatment approaches was published by Grob and colleagues (9). They were able to demonstrate that continuous daily treatment with the nsAH desloratadine resulted in significantly better quality of life as compared to on demand therapy. While these studies indicate that the treatment schedule can generally have a major impact on the outcome of treatment, the results on the efficacy of on demand nsAHs in CSU remains to be confirmed independently.

In addition to the optimal treatment schedule, there is an ongoing discussion regarding the long-term outcome of nsAH treatment. While the mode of action of nsAHs suggests a pure symptomatic therapeutic effect, there have been speculations that a disease modification effect might also occur. Indeed, in 2010, a Japanese group (Kono et al.) presented data on the EADV meeting in Gothenburg demonstrating that continuous prophylactic antihistamine therapy of CSU patients with ebastine (a nsAH) for a period of three months was associated with a lower recurrence rate after discontinuation than the same treatment lasting for only one month, provided that the drug was effective and safe during early treatment. As of yet, these results also have to be confirmed independently.

Sufficient reduction of urticarial symptoms requires higher than the licensed dosing of antihistamines in many CSU patients (10-14). In fact, increasing the dose of nsAHs up to fourfold has been shown to be more effective as compared to the standard dose in different subforms of chronic urticaria (10, 11, 14). However, for some patients even high dosed nsAHs are not enough to effectively suppress disease symptoms (11-14). The exact reasons for this are still unknown. Probably, other mediators than histamine are also involved in the development of urticaria symptoms. One such other candidate mediator is platelet activating factor (PAF). PAF is a potent phospholipid mediator with various biological activities, including platelet aggregation, airway constriction, hypotension, and vascular permeation. PAF also mediates allergic reactions and has been claimed to contribute to the pathogenesis of urticaria. Intradermal PAF injection results in a pruritic wheal and flare reaction in subjects with and without allergies (15). PAF injection is followed by a dose-dependent histamine release in vivo (16) and in cold contact urticaria, there is evidence available that PAF is an additional important mediator associated with the inflammatory reaction in the skin (17, 18). Notably, Krause et al. could demonstrate that intradermal PAF injection results in a wheal and flare type skin reaction without inducing mast cell degranulation (19). PAF may, therefore, be a relevant mediator in the pathogenesis of urticaria that acts downstream of mast cell activation and is independent of H1-receptor activation.

Rupatadine, is a drug which possesses a potent antihistamine and PAF antagonistic activity and, recently, it has been demonstrated to be safe and effective in the treatment of chronic urticaria (3, 4) and cold contact urticaria (5). Notably, it has also been shown that an increased dose of 20 mg rupatadine is more effective in the treatment of CSU symptoms as compared to the licensed 10 mg dose (20).

In summary, it seems more than reasonable to use rupatadine as a study drug in patients with CSU in order to better characterize the best nsAH treatment schedule (continuous vs. on-demand), the long-term outcome of nsAH therapy and the influence of updosing on the latter.

ELIGIBILITY:
Inclusion criteria:

* Male or female aged 18 years and older
* Documented history of active CSU (urticaria and wheals) with or without an associated angioedema for at least three days per week over the last 6 weeks prior to visit 1 (screening). Urticaria symptoms must comprise wheals and itch
* UAS7 of ≥6 during the screening phase
* Overall duration of chronic spontaneous urticaria for at least 3 months
* Informed consent signed and dated
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Willing, committed and able to return for all clinic visits and complete all study-related procedures
* In females of childbearing potential: negative pregnancy test; females willing to use highly effective contraception (Pearl-Index < 1) a woman will be considered not of childbearing potential if she is post-menopausal for > 2 years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion criteria:

* Chronic spontaneous urticaria patients with a known resistance to nsAH in 4 times the licensed doses
* Chronic spontaneous urticaria patients with a known resistance to rupatadine
* Isolated presence or domination of inducible forms of urticaria or cholinergic urticaria (no chronic spontaneous urticaria)
* History of adverse reactions to rupatadine or known hypersensitivity to rupatadine or its ingredients
* Intake of oral corticosteroids or intravenously applied corticosteroids within 28 days prior to screening visit
* Use of depot corticosteroids within 3 months prior to screening visit (inhaled corticosteroids are allowed)
* Use of systemic immunosupressants/immunomodulators such as ciclosporin, dapsone, metotrexate, and comparable drugs within 28 days prior to screening visit.
* Significant medical condition, in the opinion of the Investigator, rendering the patient immunocompromised or not suitable for a clinical trial
* Significant concomitant illness, in the opinion of the Investigator, that would adversely affect the subject's participation or evaluation in this study
* Subjects for whom there is concern, in the opinion of the Investigator, about compliance with the protocol procedures
* The presence of a permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of gastrointestinal tract)
* Presence of active cancer which requires chemotherapy or radiation therapy
* History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
* History or presence of myocardial infarction or acute myocardial ischemia
* History or presence of cardiac arrhythmia which requires drug therapy
* History or presence of clinically significant bradycardia (<50 bpm)
* ECG alterations of repolarisation (QTc prolongations >450ms in females, >430ms in males)
* Blood pressure >180/100 mmHg and/or heart rate >100/min
* Presence of uncorrected hypokalemia or hyperkalemia
* Evidence of significant hepatic or renal disease (GOT and/or GPT >2 times above the upper reference value, serum creatinine 1.5 times above the upper reference value)
* Presence of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Medication with HMG-CoA reductase inhibitors (statins)
* Presence of alcohol abuse or drug addiction
* Pregnancy or breast-feeding
* Subjects who are inmates of psychiatric wards, prisons, or other state institutions. Existing or planned placement in an institution after ruling according to § 40 passage 1, number 4 AMG (Arzneimittelgesetz).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-12; Primary Completion 2017-11-20 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Urticaria Activity Score (7 day cummulative score - UAS7) | 1 week
  The UAS daily quantifies wheals (0-3 points) and itching (0-3 points). Accordingly, the minimum and maximum value of the 7 day cumulative score (UAS7) is 0 and 42, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Allergie-Centrum-Charite, Berlin, Germany